CLINICAL TRIAL: NCT05762887
Title: Clinical Evaluation of the Antidepressant Effect of the Use of Probiotics in Bipolar Disorder and Possible Mediating Effects of Systemic and Intestinal Inflammatory Markers in the Microbiota
Brief Title: Clinical Evaluation of the Antidepressant Effect of the Use of Probiotics in Bipolar Disorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo (Other)
Collaborators: Baszucki Brain Research Fund (Other); Milken Institute (Other)
Responsible Party: Principal Investigator, Beny Lafer, Principal Investigator, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: U1111-1280-7625
Record Dates: First submitted 2023-01-11; First posted 2023-03-10 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-12

CONDITIONS: Bipolar Disorder
MeSH Terms: conditions — Bipolar Disorder

STUDY DESIGN:
Intervention Model Description: A Randomized, Double-Blind, Placebo-controlled
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All blind clinical assessments will be done by Psychiatrists, members of the University of São Paulo (USP) Bipolar Research Program managed by Michelle Flores. In this study, the intervention will be double-blind: All participants will receive the exact same pill, whether placebo or intervention, with equal packaging-manufacturing.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Probiotic group (Experimental): In addition to the usual medication treatment for bipolar disorder, following the main international guidelines for the treatment of bipolar disorder, subjects will receive food supplementation with a probiotic formulation, twice daily, with food. We will use Pendulum Therapeutics' Glucose Control, probiotic formulation patented in the United States.
  Probiotic Ingredients: Clostridium butyricum WB-STR-0006, Clostridium beijerinckii WB-STR-0005, Anaerobutyricum hallii WB-STR-0008, Akkermansia muciniphila WB-STR-0001, and Bifidobacterium infantis.
  The product also contains: Chicory inulin and oligofructose (prebiotic fiber), hypromellose (vegetarian capsule), fruit & vegetable juice (coloring agent), magnesium stearate and silica (flow agent for encapsulation)
  Interventions: Other: Probiotic Group
- Placebo Group (Placebo Comparator): In addition to the usual medication treatment for bipolar disorder, following the main international guidelines for the treatment of bipolar disorder, the subjects will receive food supplementation with a placebo formulation, twice daily, with food We will use Pendulum Therapeutics' placebo formulation that contains:
  Chicory inulin and oligofructose (prebiotic fiber), hypromellose (vegetarian capsule), fruit & vegetable juice (coloring agent), magnesium stearate and silica (flow agent for encapsulation)
  Interventions: Other: Placebo Group

INTERVENTIONS:
Other: Probiotic Group — The 84 participants will participate in a randomized, double-blind, placebo-controlled trial in two arms. The probiotic group will consist of 42 patients. These patients will be recruited from the USP Bipolar Disorder Program. This program has an outpatient clinic that offers free medical care to a population of different ethnic groups, with the majority of subjects coming from the middle and lower social classes.
  Arms: Probiotic group
Other: Placebo Group — The 84 participants will participate in a randomized, double-blind, placebo-controlled trial in two arms. The placebo group will consist of 42 patients. These patients will be recruited from the USP Bipolar Disorder Program. This program has an outpatient clinic that offers free medical care to a population of different ethnic groups, with the majority of subjects coming from the middle and lower social classes.
  Arms: Placebo Group

SUMMARY:
Bipolar Disorder (BD) is highly incapacitating and associated with premature mortality. Depressive symptoms and episodes are the most frequent cause of disability in subjects with BD and over half of patients do not respond adequately to approved treatments for this condition, showing the need for new classes of treatments to complement current pharmacotherapy. Previous studies demonstrated that the intestinal flora have potential positive or negative effects on the Central Nervous System and suggest that adding specific strains of bacteria to people's diet may have antidepressant properties.The study proposes to evaluate the clinical benefit of adding probiotics to pharmacological treatments for bipolar depression. This will be a study with 84 subjects (42 receiving probiotics and 42 placebo). The research team in this department has focused especially on non-pharmacological treatments for bipolar disorder (psychotherapy, nutrition and exercise) and is multidisciplinary in scope with psychiatrists, psychologists, nurses, physiotherapists and nutritionists participating in research projects.

DETAILED DESCRIPTION:
It will test, in a proof-of-concept study, the antidepressant efficacy of adjunctive administration of probiotics in bipolar depression and evaluate potential inflammatory and metabolic markers associated with response to treatment. With this objective, 84 individuals with bipolar disorder type I or type II presenting subsyndromal depressive symptoms or a major depressive episode will be recruited. The study design lasts 12 weeks and is expected to last two years.

ELIGIBILITY:
Inclusion Criteria:

* BD type I or type II, according to the use of Mini Internacional Neuropsychiatric Interview (MINI)
* Score on the Young Mania Rating Scale (YMRS) < 8
* Score on the Montgomery-Asberg Depression Rating Scale (MADRS) > 8
* Be receiving major guideline-approved treatments for bipolar depression for at least 4 weeks

Exclusion Criteria:

* Pregnant or lactating women
* Substance or alcohol dependence
* Patients on prolonged antibiotic therapy, immunosuppressive therapies
* A recent introduction of antidepressants in the last 15 days
* Use of another probiotic, either in the form of food, sachets, capsules and others

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2023-01-09 (Actual); Primary Completion 2024-08-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Outcome | 12 weeks
  The Montgomery-Asberg Depression Rating Scale (MADRS) will be used in order to evaluate the reduction of depressive symptoms. Response to treatment at week-12 will be defined as ≥ 50% reduction in total MADRS total score from baseline. Remission will be defined as MADRS total score ≤ 12.

CONTACTS AND LOCATIONS:
Overall Officials: Beny lafer, PhD, Principal Investigator — University of Sao Paulo
Locations (1):
- University of Sao Paulo, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ho P, Ross DA. More Than a Gut Feeling: The Implications of the Gut Microbiota in Psychiatry. Biol Psychiatry. 2017 Mar 1;81(5):e35-e37. doi: 10.1016/j.biopsych.2016.12.018. No abstract available. PMID 28137375
- [Result] Dinan TG, Cryan JF. The Microbiome-Gut-Brain Axis in Health and Disease. Gastroenterol Clin North Am. 2017 Mar;46(1):77-89. doi: 10.1016/j.gtc.2016.09.007. Epub 2017 Jan 4. PMID 28164854
- [Result] Huang R, Wang K, Hu J. Effect of Probiotics on Depression: A Systematic Review and Meta-Analysis of Randomized Controlled Trials. Nutrients. 2016 Aug 6;8(8):483. doi: 10.3390/nu8080483. PMID 27509521
- [Result] Miyaoka T, Kanayama M, Wake R, Hashioka S, Hayashida M, Nagahama M, Okazaki S, Yamashita S, Miura S, Miki H, Matsuda H, Koike M, Izuhara M, Araki T, Tsuchie K, Azis IA, Arauchi R, Abdullah RA, Oh-Nishi A, Horiguchi J. Clostridium butyricum MIYAIRI 588 as Adjunctive Therapy for Treatment-Resistant Major Depressive Disorder: A Prospective Open-Label Trial. Clin Neuropharmacol. 2018 Sep/Oct;41(5):151-155. doi: 10.1097/WNF.0000000000000299. PMID 30234616
- [Result] Perraudeau F, McMurdie P, Bullard J, Cheng A, Cutcliffe C, Deo A, Eid J, Gines J, Iyer M, Justice N, Loo WT, Nemchek M, Schicklberger M, Souza M, Stoneburner B, Tyagi S, Kolterman O. Improvements to postprandial glucose control in subjects with type 2 diabetes: a multicenter, double blind, randomized placebo-controlled trial of a novel probiotic formulation. BMJ Open Diabetes Res Care. 2020 Jul;8(1):e001319. doi: 10.1136/bmjdrc-2020-001319. PMID 32675291
- [Result] Yatham LN, Kennedy SH, Parikh SV, Schaffer A, Bond DJ, Frey BN, Sharma V, Goldstein BI, Rej S, Beaulieu S, Alda M, MacQueen G, Milev RV, Ravindran A, O'Donovan C, McIntosh D, Lam RW, Vazquez G, Kapczinski F, McIntyre RS, Kozicky J, Kanba S, Lafer B, Suppes T, Calabrese JR, Vieta E, Malhi G, Post RM, Berk M. Canadian Network for Mood and Anxiety Treatments (CANMAT) and International Society for Bipolar Disorders (ISBD) 2018 guidelines for the management of patients with bipolar disorder. Bipolar Disord. 2018 Mar;20(2):97-170. doi: 10.1111/bdi.12609. Epub 2018 Mar 14. PMID 29536616